CLINICAL TRIAL: NCT04621084
Title: Influence of the COVId-19 Pandemic on STRESS and Eating Habits
Acronym: COVISTRESSNutr
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2020 COVISTRESS NUTRITION
Record Dates: First submitted 2020-11-05; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Nutrition
Keywords: nutrition; Covid-19; Eating habits; Stress
MeSH Terms: conditions — COVID-19; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Eating habits — Questionnary online

SUMMARY:
The Coronavirus has caused containment of more than a third of the world's population. Containment can drastically change lifestyle habits, including eating habits such as the number of meals, meal times or their composition. However, there is currently no data on the influence of confinement on eating habits.

DETAILED DESCRIPTION:
This is an observational study by REDCap questionnaire® via a flyer deposited in the waiting room of the COVID screening centres. No incentive to complete the questionnaire will be made.

The self-administered questionnaire will assess stress, changes in eating habits, and relationships with socio-demographic or lifestyle factors.

This questionnaire includes 9 specific questions on nutrition and 40 general questions.

ELIGIBILITY:
Inclusion Criteria:

* All volunteers who are screened

Exclusion Criteria:

* none

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All volunteers
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Stress measures | Day 1
  Attitudes and stress related to screening procedure will be measured via questionnaire

SECONDARY OUTCOMES:
Nutrition | Day 1
  Eating habits will be measured via questionnaire

OTHER OUTCOMES:
Sociodemographic characteristics | Day 1
  Age, gender, qualification, personal work status, ethnicity, life characteristics and stress will be assessed by questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, AURA, France